CLINICAL TRIAL: NCT06551415
Title: Dabigatran Versus Apixaban in Cerebral Venous Thrombosis, a Randomized Controlled Trial
Brief Title: Dabigatran Versus Apixaban in Cerebral Venous Thrombosis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Mohamed G. zeinhom, MD, principal investigator, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2309088
Record Dates: First submitted 2024-08-09; First posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Cerebral Venous Sinus Thrombosis
Keywords: apixaban,; cerebral venous thrombosis; Dabigatran; Egypt
MeSH Terms: conditions — Intracranial Thrombosis | interventions — Dabigatran; apixaban

STUDY DESIGN:
Intervention Model Description: We compared the efficacy and safety of a Dabigatran 150 mg Bid administered within 24 hours of randomization after having first-ever cerebral venous thrombosis compared to apixaban 5mg Bid were assessed through rate of recurrent VTE, mRS, rate of venous recanalization, HIT score, MoCA test, and central and peripheral hemorrhagic complications
Who Masked: Investigator, Outcomes Assessor
Masking Description: An independent statistician generated a blocked randomization sequence using computer-generated random numbers; in a one-to-one ratio, participants were randomly assigned to receive doses of Dabigatran or rivaroxaban by a specially trained and qualified nurse. We prepared Sequentially numbered opaque sealed envelopes and 580 labels for each drug labeled Drug A or B. According to the randomization chart, put them into envelopes numbered 1 to 580. Envelopes were attached to the patient's files. Patients were recruited sequentially and were given enrollment numbers starting from 1, which were mentioned in their files. Files with the same number as the patient enrolment number were opened, and the patients were assigned to receive drugs A or B. Drug A included dabigatran, and Drug B included apixaban. The statistical analysis was performed by an independent statistician who did not know the treatment protocol of groups A or B.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dabigatran (Active Comparator): 100 CVT patients will receive dabigatran 150mg Bid for 6 months. We will assess the Proportion of subjects who have partial or complete venous recanalization by Day 180 the rate of drug hemorrhagic complications using the PLATO bleeding definition, and the rates of patients who achieved a favorable outcome with (mRS = 0-2) after one week and after 180 days in a face-to-face interview in the outpatient clinic, Proportion of subjects with recurrent venous thromboembolism (any thrombosis at a new site, including cerebral venous thrombosis in a separate location from the index event) at Day 180 or the end of anticoagulation, whichever is sooner, rates of a composite of pulmonary embolism, DVT, myocardial infarction, and death due to vascular events after 180 days of follow-up, the MoCA, HIT-6 by 180 days, the rate of treatment-related adverse effects assessed by a follow-up questionnaire
  Interventions: Drug: Dabigatran Etexilate 150mg
- apixaban (Active Comparator): 100 CVT patients will receive apixaban 5mg Bid for 6 months. We will assess the Proportion of subjects who have partial or complete venous recanalization by Day 180 the rate of drug hemorrhagic complications using the PLATO bleeding definition, and the rates of patients who achieved a favorable outcome with (mRS = 0-2) after one week and after 180 days in a face-to-face interview in the outpatient clinic, Proportion of subjects with recurrent venous thromboembolism (any thrombosis at a new site, including cerebral venous thrombosis in a separate location from the index event) at Day 180 or the end of anticoagulation, whichever is sooner, rates of a composite of pulmonary embolism, DVT, myocardial infarction, and death due to vascular events after 180 days of follow-up, the MoCA, HIT-6 by 180 days, the rate of treatment-related adverse effects assessed by a follow-up questionnaire
  Interventions: Drug: Apixaban 5MG

INTERVENTIONS:
Drug: Dabigatran Etexilate 150mg — 100 CVT patients will receive dabigatran 150mg Bid for 6 months. We will assess the Proportion of subjects who have partial or complete venous recanalization by Day 180 the rate of drug hemorrhagic complications using the PLATO bleeding definition, and the rates of patients who achieved a favorable outcome with (mRS = 0-2) after one week and after 180 days in a face-to-face interview in the outpatient clinic, Proportion of subjects with recurrent venous thromboembolism (any thrombosis at a new site, including cerebral venous thrombosis in a separate location from the index event) at Day 180 or the end of anticoagulation, whichever is sooner, rates of a composite of pulmonary embolism, DVT, myocardial infarction, and death due to vascular events after 180 days of follow-up, the MoCA, HIT-6 by 180 days, the rate of treatment-related adverse effects assessed by a follow-up questionnaire
  Other Names: group A
  Arms: Dabigatran
Drug: Apixaban 5MG — 100 CVT patients will receive apixaban 5mg Bid for 6 months. We will assess the Proportion of subjects who have partial or complete venous recanalization by Day 180 the rate of drug hemorrhagic complications using the PLATO bleeding definition, and the rates of patients who achieved a favorable outcome with (mRS = 0-2) after one week and after 180 days in a face-to-face interview in the outpatient clinic, Proportion of subjects with recurrent venous thromboembolism (any thrombosis at a new site, including cerebral venous thrombosis in a separate location from the index event) at Day 180 or the end of anticoagulation, whichever is sooner, rates of a composite of pulmonary embolism, DVT, myocardial infarction, and death due to vascular events after 180 days of follow-up, the MoCA, HIT-6 by 180 days, the rate of treatment-related adverse effects assessed by a follow-up questionnaire.
  Other Names: group B
  Arms: apixaban

SUMMARY:
Along with the current clinical trial, the efficacy and safety of a 150 mg Bid dabigatran administered within 24 hours of randomization after having first-ever cerebral venous thrombosis compared to apixaban 5mg Bid were assessed through rate of recurrent VTE, mRS, rate of venous recanalization, HIT score, MoCA test, and central and peripheral hemorrhagic complications

DETAILED DESCRIPTION:
The investigators conducted a single-blinded randomized controlled trial between August 2021 and August 2024 after the ethics committee of the faculty of medicine at Kafr el-Sheik University approved it.

The investigators got written informed consent from all eligible patients or their first order of kin before randomization.

The study will be composed of 2 arms Dabigatran arm, which consisted of 100 patients who received 150 mg Bid dabigatran daily for 6 months, and the apixaban arm, consisting of 100 patients who received (5 mg Bid for 6 months),

Study Procedures:

Every patient in our study will undergo:

Clinical workup: History, clinical assessment, NIHSS, MoCA, HIT-6, and mRS were recorded at baseline and 30,90,180 days as a follow-up.

Detection of Risk Factors & Profiles:

Echocardiography TTE: in indicated patients ECG Monitoring: daily ECG monitoring will be performed in indicated patients. 3- Carotid Duplex: carotid duplex in indicated patients.

4- ESR & Lipid Profile& liver functions: All will be tested routinely for all patients.

5- Non-contrast CT brain and CTV on admission or MRI and MRV:, at baseline and after 6 months of treatment CT brain: Any patient with unexplained clinical deterioration at any time throughout his/her hospital stay will be urgently imaged by CT.

Primary End Point:

The primary efficacy outcome was the rate of Proportion of subjects with partial or complete venous recanalization by Day 180, and the primary safety outcome was the rate of drug hemorrhagic complications using the PLATO bleeding definition.

• Secondary End Point: The secondary efficacy outcomes were to evaluate the rates of patients who achieved a favorable outcome with (mRS = 0-2) after one week and after 180 days in a face-to-face interview in the outpatient clinic, Proportion of subjects with recurrent venous thromboembolism (any thrombosis at a new site, including cerebral venous thrombosis in a separate location from the index event) at Day 180 or the end of anticoagulation, whichever is sooner, rates of a composite of pulmonary embolism, DVT, myocardial infarction, and death due to vascular events after 180 days of follow-up, the MoCA, HIT-6 by 180 days, while the secondary safety outcome was the rate of treatment-related adverse effects assessed by a follow-up questionnaire

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 and above
2. New diagnosis of symptomatic cerebral venous thrombosis as confirmed on CT/CT venogram or MRI/MR venogram
3. Ability to randomize within 14 days of neuroimaging-confirmed diagnosis
4. The treating clinician thinks that the patient is appropriate for oral anticoagulation as per the standard of care
5. The patient or legally authorized representative can give written informed consent

Exclusion Criteria:

1. The patient has known antiphospholipid antibody syndrome with a previous history of venous or arterial thrombosis
2. The patient is anticipated to require invasive procedures (e.g., lumbar puncture, thrombectomy, hemicraniectomy) before initiation of oral anticoagulation
3. Patient is unable to swallow due to a depressed level of consciousness
4. Impaired renal function (i.e., CrCl < 30 mL/min using CockroftGault equation)
5. Pregnancy: if a woman is of childbearing potential, a urine or serum beta-human chorionic gonadotropin (β-hCG) test is positive
6. Breastfeeding at the time of randomization
7. Bleeding diathesis or other contraindication to anticoagulation
8. Any concurrent medical condition requiring mandatory antiplatelet or anticoagulant use
9. Concomitant use of strong CYP3A4 inducers (e.g., ongoing use of Dilantin, carbamazepine, HIV protease inhibitors) or CYP3A4 inhibitors (e.g., diltiazem, ketoconazole)
10. The patient has a severe or fatal comorbid illness that will prevent improvement

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects who have partial or complete venous recanalization by Day 180 | 180 days
  The investigators will perform magnetic resonance venography for all patients after 6 months to show if there is partial or complete recanalization of the affected venous sinus
Rate of drug-related hemorrhagic complications | 180 days
  the rate of drug hemorrhagic complications which was evaluated using the PLATO bleeding definition which classified hemorrhagic complications into three types as follows: Major bleeding which had one or more of the following criteria: fatal bleeding, intracranial, intrapericardial, bleeding associated with reduction of hemoglobin > 3-5 g/dl, bleeding required transfusion of two to four units whole blood or PRBCs, bleeding produced hypovolemic shock or severe hypotension that required pressor or surgery; Minor bleeding that required medical intervention to stop or treat bleeding: Minimal bleeding: any bleeding that did not require intervention or treatment such as bruising, bleeding gums, oozing from injection sites.

SECONDARY OUTCOMES:
value of Modified Rankin Scale (mRS) at six months | 6 months
  mRS measures the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. Its value ranges from 0 to 6; the lower the score, the better the stroke outcome. A favorable stroke outcome is considered with an mRS value equal to two or less.
value of HIT-6 score in each group after six months of treatment | 6 months
  The investigators assessed the absolute change in HIT6 score, the Headache Impact Test-6 (HIT-6) assessed the burden of headache in each group; the HIT-6 consists of six items: pain, social functioning, role functioning, vitality, cognitive functioning, and psychological distress, the patient answers each of the six related questions using one of the following five responses: "never", "rarely", "sometimes", "very often," or "always." These responses are summed to produce a total HIT-6 score that ranges from 36 to 78, where a higher score indicates a greater impact of headache on the daily life of the respondent. It has four impact grades: little-to-no impact (HIT-6 score: 36-49), moderate impact (HIT-6 score: 50-55), substantial impact (HIT-6 score: 56-59), and severe impact (HIT-6 score: 60-78)
rate of drug adverse effects | 6 months
  Drug adverse effects: all non-hemorrhagic side effects related to the drugs of our study will be reported
The proportion of participants with recurrent venous thromboembolism | 6 months
  The investigators will assess the proportion of participants with recurrent venous thromboembolism (any thrombosis at a new site, including CVT in a separate location from the index event) during 6 months of treatment
rate of composite pulmonary embolism, myocardial infarction, and death due to vascular events | 6 months
  The investigators will assess the proportion of participants with pulmonary embolism, myocardial infarction, and death due to vascular events at during 6 months of treatment

CONTACTS AND LOCATIONS:
Overall Officials: mohamed G. Zeinhom, MD, Principal Investigator — neurology department kafr el-sheikh university
Locations (1):
- Kafr Elsheikh University Hospital, Kafr ash Shaykh, Egypt

IPD SHARING:
Plan to Share IPD: No
All the data supporting this research's findings will be available from the corresponding author, Dr. Mohamed G. Zeinhom, upon reasonable request.

REFERENCES:
- [Result] Paciaroni M, Ince B, Hu B, Jeng JS, Kutluk K, Liu L, Lou M, Parfenov V, Wong KSL, Zamani B, Paek D, Min Han J, Del Aguila M, Girotra S. Benefits and Risks of Clopidogrel vs. Aspirin Monotherapy after Recent Ischemic Stroke: A Systematic Review and Meta-Analysis. Cardiovasc Ther. 2019 Dec 1;2019:1607181. doi: 10.1155/2019/1607181. eCollection 2019. PMID 31867054
- [Result] Meyer DM, Albright KC, Allison TA, Grotta JC. LOAD: a pilot study of the safety of loading of aspirin and clopidogrel in acute ischemic stroke and transient ischemic attack. J Stroke Cerebrovasc Dis. 2008 Jan-Feb;17(1):26-9. doi: 10.1016/j.jstrokecerebrovasdis.2007.09.006. PMID 18190818